CLINICAL TRIAL: NCT03363321
Title: A MULTICENTER, OPEN-LABEL STUDY TO EVALUATE THE LONG-TERM SAFETY, TOLERABILITY AND EFFICACY OF SUBCUTANEOUS PF-06741086 IN SUBJECTS WITH SEVERE HEMOPHILIA
Brief Title: PF-06741086 Long-term Treatment in Severe Hemophilia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: B7841003; 2017-001255-31 (EudraCT Number)
Record Dates: First submitted 2017-11-30; First posted 2017-12-06 (Actual); Results first posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Hemophilia A or B
Keywords: hemophilia
MeSH Terms: conditions — Hemophilia A | interventions — marstacimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- PF-06741086 (Cohort 1) (Experimental)
  Interventions: Biological: PF-06741086
- PF-06741086 (Cohort 2) (Experimental)
  Interventions: Biological: PF-06741086
- PF-06741086 (Cohort 3) (Experimental)
  Interventions: Biological: PF-06741086
- PF-06741086 (Cohort 4) (Experimental)
  Interventions: Biological: PF-06741086
- PF-06741086 (Cohort 5) (Experimental)
  Interventions: Biological: PF-06741086
- PF-06741086 (Cohort 6) (Experimental)
  Interventions: Biological: PF-06741086

INTERVENTIONS:
Biological: PF-06741086 — PF-06741086 subcutaneous injection

SUMMARY:
This study is designed to evaluate the safety, tolerability and efficacy of long-term treatment with PF-06741086 in subjects with severe hemophilia who participated in the 3-month Phase 1b/2 B7841002 study. Additionally, de novo subjects will be recruited into this study.

ELIGIBILITY:
Inclusion Criteria:

* Severe hemophilia A or B (Factor VIII or Factor IX activity ≤ 1%)
* Subjects enrolled as Factor VIII or Factor IX inhibitor patients must have a positive inhibitor test result (above the upper limit of normal) at the local laboratory and must receive a bypass agent as primary treatment for bleeding episodes.
* Episodic (on-demand) treatment regimen prior to screening
* At least 6 acute bleeding episodes during the 6-month period prior to screening

Exclusion Criteria:

* Known coronary artery, thrombotic, or ischemic disease
* Concomitant treatment with activated prothrombin complex concentrate

Ages: 12 Years to 74 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2020-08-05 (Actual); Study Completion 2020-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- UC Denver Hemophilia and Thrombosis Center, Aurora, Colorado, United States
- Centro de Hematologia e Hemoterapia de Campinas- Hemocentro de Campinas, Campinas, São Paulo, Brazil
- Hospital Dr. Sotero del Rio, Santiago, Puente ALTO, Chile
- Klinicki bolnicki centar Zagreb, Zagreb, Croatia
- Klinika Hematologii i Transplantologii Uniwersyteckie Centrum Kliniczne, Gdansk, Poland
- South Africa (2):
  - Phoenix Pharma (Pty) Ltd, Port Elizabeth, Eastern Cape
  - Charlotte Maxeke Johannesburg Academic Hospital, Johannesburg, Gauteng
- UniversitatsSpital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Mahlangu J, Luis Lamas J, Cristobal Morales J, Malan DR, Teeter J, Charnigo RJ, Hwang E, Arkin S. Long-term safety and efficacy of the anti-tissue factor pathway inhibitor marstacimab in participants with severe haemophilia: Phase II study results. Br J Haematol. 2023 Jan;200(2):240-248. doi: 10.1111/bjh.18495. Epub 2022 Oct 11. PMID 36220152
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7841003

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twenty-four participants were screened, of which, 4 failed at screening. All the 20 participants who met the eligibility criteria were assigned to the study treatment and were treated with marstacimab. Among 20 participants treated with marstacimab, 18 completed the study, and 2 discontinued from study due to withdrawal by participant, which were not related to safety.
Groups:
- Cohort 1: 300mg - 300mg Non-Inhibitor: Participants without inhibitors to Factor VIII (FVIII) or Factor IX (FIX) from Cohort 1 of Study 1002 (B7841002, NCT02974855) continued to receive PF-06741086 300 mg subcutaneously (SC) once weekly (QW) from Day 1 to Day 365.
- Cohort 2: 300mg Loading + 150mg - 300mg Loading + 150mg Non-Inhibitor: Participants without inhibitors to FVIII or FIX from Cohort 2 of Study 1002 continued to receive PF-06741086 300 mg loading dose on Day 1 and 150 mg SC QW from Day 29 to Day 365.
- Cohort 3: 450mg - 300mg Loading + 150mg Non-Inhibitor: Participants without inhibitors to FVIII or FIX from Cohort 3 (450 mg SC) of Study 1002 started to receive PF-06741086 300 mg loading dose on Day 1 and 150 mg SC QW from Day 29 to Day 365.
- Cohort 4: 300mg - 300mg Inhibitor: Participants with inhibitors to FVIII or FIX from Cohort 4 (300 mg SC) of Study 1002 continued to receive PF-06741086 300 mg SC QW from Day 1 to Day 365.
- Cohort 5: De Novo 300mg Loading + 150mg Inhibitors: De Novo participants with inhibitors to FVIII or FIX received a 300 mg SC loading dose on Day 1, and then followed by 150 mg SC QW to Day 365.
Period: Overall Study
Arm/Group | Cohort 1: 300mg - 300mg Non-Inhibitor | Cohort 2: 300mg Loading + 150mg - 300mg Loading + 150mg Non-Inhibitor | Cohort 3: 450mg - 300mg Loading + 150mg Non-Inhibitor | Cohort 4: 300mg - 300mg Inhibitor | Cohort 5: De Novo 300mg Loading + 150mg Inhibitors
Started | 5 | 4 | 4 | 5 | 2
Completed | 5 | 3 | 4 | 4 | 2
Not Completed | 0 | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants who received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: 300mg - 300mg Non-Inhibitor | Cohort 2: 300mg Loading + 150mg - 300mg Loading + 150mg Non-Inhibitor | Cohort 3: 450mg - 300mg Loading + 150mg Non-Inhibitor | Cohort 4: 300mg - 300mg Inhibitor | Cohort 5: De Novo 300mg Loading + 150mg Inhibitors | Total
Number analyzed (Participants) | 5 | 4 | 4 | 5 | 2 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 4 | 5 | 2 | 20
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.0 (9.70) | 31.3 (10.63) | 41.8 (16.24) | 42.0 (5.24) | 20.0 (1.41) | 35.4 (11.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 5 | 4 | 4 | 5 | 2 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 1 | 1 | 0 | 7
  Not Hispanic or Latino | 2 | 2 | 3 | 4 | 2 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 0 | 2 | 0 | 6
  White | 3 | 2 | 4 | 3 | 2 | 14
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), TEAEs by Severity, and Serious Adverse Events (SAEs) (All Causality and Treatment-Related)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a product; the event did not need to have a causal relationship with the treatment. A serious adverse event (SAE) was any untoward medical occurrence at any dose that resulted in death; was life threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth defect. AEs included both SAEs and non-serious AEs. TEAEs were AEs occurred following the start of treatment or AEs increasing in severity during treatment. Treatment-related TEAEs were determined by the investigator. Grades 3 AEs were severe and undesirable adverse events. Grades 4 AEs were life threatening or disabling adverse events.
Time Frame: Day 1 up to Day 393
Population: The analysis population included all participants who received at least 1 dose of investigational product. Here "Overall Number of Participants Analyzed" signifies number of participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: 300mg - 300mg Non-Inhibitor | Cohort 2: 300mg Loading + 150mg - 300mg Loading + 150mg Non-Inhibitor | Cohort 3: 450mg - 300mg Loading + 150mg Non-Inhibitor | Cohort 4: 300mg - 300mg Inhibitor | Cohort 5: De Novo 300mg Loading + 150mg Inhibitors
Number analyzed (Participants) | 5 | 4 | 4 | 5 | 2
Participants
  All-causalities TEAE | 5 | 2 | 4 | 2 | 1
  Treatment-related TEAE | 2 | 0 | 0 | 0 | 1
  All-causalities serious TEAE | 1 | 0 | 0 | 0 | 0
  Treatment-related serious TEAE | 0 | 0 | 0 | 0 | 0
  All-causalities Grade 3 or 4 TEAE | 1 | 0 | 0 | 0 | 1
  Treatment-related Grade 3 or 4 TEAE | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Abnormal Laboratory Findings Without Regard to Baseline Abnormality (Including Hematology, Serum Chemistry, and Urinalysis)
Description: Following parameters were analyzed for laboratory examination: hematology, clinical chemistry, and urinalysis. The hematology parameters and pre-defined criteria included: neutrophils (10^3/millimeter[mm]^3) <0.8*lower limit of normal (LLN), and basophils (10^3/mm^3) >1.2*upper limit of normal (ULN). The clinical chemistry parameter and pre-defined criteria included: bilirubin (milligrams [mg]/decilitre [dL]) >1.5 ULN, aspartate aminotransferase (units [U]/liter [L]) >3.0 ULN, glucose (mg/dL) >1.5*ULN. The urinalysis parameter and pre-defined criteria included: urine glucose ≥1, ketones (scalar) ≥1, urine protein ≥1, urine hemoglobin (scalar) ≥1, and hyaline casts per low power field (/LPF). Participants met criteria at any time point were included.
Time Frame: Hematology and serum chemistry: Baseline, Days 1, 29, 57, 85, 169, 253, and 365 visits. Urinalysis: Baseline, Days 1, 85, 169, 253, and 365 visits.
Population: This analysis population included all participants who received at least 1 dose of investigational product. Here "Overall Number of Participants Analyzed" signifies number of participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: 300mg - 300mg Non-Inhibitor | Cohort 2: 300mg Loading + 150mg - 300mg Loading + 150mg Non-Inhibitor | Cohort 3: 450mg - 300mg Loading + 150mg Non-Inhibitor | Cohort 4: 300mg - 300mg Inhibitor | Cohort 5: De Novo 300mg Loading + 150mg Inhibitors
Number analyzed (Participants) | 5 | 3 | 4 | 5 | 2
Participants
  Hematology Neutrophils (10^3/mm^3) <0.8*LLN | 1 | 1 | 0 | 0 | 0
  Hematology Basophils (10^3/mm^3) >1.2*ULN | 0 | 0 | 0 | 1 | 1
  Clinical Chemistry Bilirubin (mg/dL) >1.5*ULN | 0 | 0 | 0 | 0 | 1
  Clinical Chemistry Aspartate Aminotransferase (U/L) >3.0*ULN | 0 | 0 | 0 | 0 | 1
  Clinical Chemistry Glucose (mg/dL) >1.5*ULN | 0 | 0 | 1 | 1 | 0
  Urinalysis URINE Glucose ≥1 | 0 | 0 | 1 | 0 | 0
  Urinalysis Ketones (Scalar) ≥1 | 1 | 0 | 0 | 0 | 0
  Urinalysis URINE Protein ≥1 | 0 | 1 | 0 | 0 | 0
  Urinalysis URINE Hemoglobin (Scalar) ≥1 | 0 | 0 | 1 | 0 | 0
  Urinalysis Hyaline Casts (/LPF) >1: number analyzed (Participants) | 0 | 1 | 0 | 1 | 1
  Urinalysis Hyaline Casts (/LPF) >1 | 0 | 1 | 0 | 1 | 0

3. Primary Outcome: Number of Participants With Changes From Baseline in Vital Signs Measurements Meeting the Pre-Defined Categorical Summarization Criteria
Description: Following parameters were analyzed for vital sign examination: blood pressure (BP), pulse rate (PR), temperature, respiration rate. Categorical vital signs: Temperature >38.5 degree(s) Celsius (℃), Supine PR: <40 or >120 beats per minute (BPM), Systolic BP: <90 mm Hg, >=30 mm Hg change from baseline, Diastolic BP: <50 mm Hg, >=20 mm Hg change from baseline.
Time Frame: Baseline, Days 1, 29, 57, 85, 113, 141, 169, 197, 225, 253, 281, 309, 337, 365 and 393 visits.
Population: This analysis population included all participants who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: 300mg - 300mg Non-Inhibitor | Cohort 2: 300mg Loading + 150mg - 300mg Loading + 150mg Non-Inhibitor | Cohort 3: 450mg - 300mg Loading + 150mg Non-Inhibitor | Cohort 4: 300mg - 300mg Inhibitor | Cohort 5: De Novo 300mg Loading + 150mg Inhibitors
Number analyzed (Participants) | 5 | 4 | 4 | 5 | 2
Participants
  Systolic BP (mmHg) < 90 | 0 | 0 | 0 | 0 | 0
  Systolic BP Change ≥30 mm Hg increase | 0 | 0 | 1 | 0 | 0
  Systolic BP Change ≥30 mm Hg decrease | 0 | 1 | 0 | 1 | 0
  Diastolic BP (mmHg) < 50 | 0 | 0 | 0 | 0 | 0
  Diastolic BP Change ≥20 mm Hg increase | 1 | 0 | 1 | 1 | 0
  Diastolic BP Change ≥20 mm Hg decrease | 0 | 1 | 1 | 1 | 0
  Supine PR (BPM) <40 | 0 | 0 | 0 | 0 | 0
  Supine PR (BPM) >120 | 0 | 0 | 0 | 0 | 0
  Temperature >38.5 ℃ | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Change From Baseline in Electrocardiogram (ECG) Parameters Meeting the Pre-defined Categorical Summarization Criteria
Description: Baseline was defined as the average of triplicate ECG measurements collected prior to dosing on Day 1 in B7841003. Criteria for potentially clinically important changes in ECG were defined as: PR interval value >=300 millisecond (msec); PR interval baseline >200 msec and change >=25%; PR interval baseline <=200 msec and change >=50%; QRS complex value >=140 msec and change >=50%; QTcF value >=450 msec and change >=30 msec. Only the number of participants meeting pre-defined criteria was reported below.
Time Frame: Baseline, Days 1 and 29 visits
Population: ECG was only evaluated in de novo participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 5: De Novo 300mg Loading + 150mg Inhibitors
Number analyzed (Participants) | 2
Participants
  PR interval value >=300 msec | 0
  PR interval baseline >200 msec and Change >=25% | 0
  PR interval baseline <=200 msec and change >=50% | 0
  QRS complex value >=140 msec | 0
  QRS complex change >=50% | 0
  450 <= QTcF Value (msec) < 480 | 0
  480 <= QTcF Value (msec) < 450 | 0
  QTcF Value >= 500 msec | 0
  30 <= QTcF Change (msec) < 60 | 0
  QTcF Change >= 60 msec | 0

5. Primary Outcome: Number of Participants With Abnormalities in Physical Examination Findings
Description: Physical examinations were conducted by a physician, trained physician's assistant, or nurse practitioner as acceptable according to local regulation. A full physical examination included head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, gastrointestinal, musculoskeletal, and neurological systems. The limited or abbreviated physical examination was focused on general appearance, the respiratory and cardiovascular systems, as well as towards participant reported symptoms. For measuring weight, a scale with appropriate range and resolution was used and must have been placed on a stable, flat surface. Participants removed shoes, bulky layers of clothing, and jackets so that only light clothing remains. They also removed the contents of their pockets and remain still during measurement of weight.
Time Frame: Day 1 to Day 393
Population: The analysis population included all participants who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: 300mg - 300mg Non-Inhibitor | Cohort 2: 300mg Loading + 150mg - 300mg Loading + 150mg Non-Inhibitor | Cohort 3: 450mg - 300mg Loading + 150mg Non-Inhibitor | Cohort 4: 300mg - 300mg Inhibitor | Cohort 5: De Novo 300mg Loading + 150mg Inhibitors
Number analyzed (Participants) | 5 | 4 | 4 | 5 | 2
Participants | 5 | 2 | 3 | 4 | 2

6. Primary Outcome: Number of Participants With Injection Site Reactions
Description: Injection site reactions included but were not limited to: erythema, induration, ecchymosis, pain and pruritus. Grade of severity was defined as follows: Mild: Transient or mild discomfort (< 48 hours); no medical intervention/therapy required. Moderate: Mild to moderate limitation in activity - some assistance may be needed; no or minimal medical intervention/therapy required. Severe: Marked limitation in activity, some assistance usually required; medical intervention/therapy required, hospitalizations possible.
Time Frame: Day 1 to Day 365, and Day 393 visit.
Population: This analysis population included all participants who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: 300mg - 300mg Non-Inhibitor | Cohort 2: 300mg Loading + 150mg - 300mg Loading + 150mg Non-Inhibitor | Cohort 3: 450mg - 300mg Loading + 150mg Non-Inhibitor | Cohort 4: 300mg - 300mg Inhibitor | Cohort 5: De Novo 300mg Loading + 150mg Inhibitors
Number analyzed (Participants) | 5 | 4 | 4 | 5 | 2
Participants
  Erythema (redness) Mild | 0 | 0 | 0 | 0 | 0
  Erythema (redness) Moderate | 0 | 0 | 0 | 0 | 0
  Erythema (redness) Severe | 0 | 0 | 0 | 0 | 1
  Induration (swelling) Mild | 1 | 0 | 0 | 0 | 0
  Induration (swelling) Moderate | 0 | 0 | 0 | 0 | 0
  Induration (swelling) Severe | 0 | 0 | 0 | 0 | 1
  Ecchymosis (bruising) Mild | 1 | 0 | 0 | 0 | 0
  Ecchymosis (bruising) Moderate | 0 | 0 | 0 | 0 | 0
  Ecchymosis (bruising) Severe | 0 | 0 | 0 | 0 | 0
  Pain (after injection) Mild | 1 | 0 | 0 | 0 | 0
  Pain (after injection) Moderate | 0 | 0 | 0 | 0 | 0
  Pain (after injection) Severe | 0 | 0 | 0 | 0 | 0
  Pruritus (itching) Mild | 1 | 0 | 0 | 0 | 0
  Pruritus (itching) Moderate | 0 | 0 | 0 | 0 | 0
  Pruritus (itching) Severe | 0 | 0 | 0 | 0 | 0
  Other Mild | 1 | 0 | 0 | 0 | 0
  Other Moderate | 0 | 0 | 0 | 0 | 0
  Other Severe | 0 | 0 | 0 | 0 | 1
  Any injection site reaction Mild | 2 | 0 | 0 | 0 | 0
  Any injection site reaction Moderate | 0 | 0 | 0 | 0 | 0
  Any injection site reaction Severe | 0 | 0 | 0 | 0 | 1

7. Secondary Outcome: Annualized Bleeding Rate (ABR)
Description: The ABR was calculated as ([number of bleeding events × 365.25] / observed treatment period in days)
Time Frame: Day 1 to Day 365, and Day 393 visit. Pre-Treatment summarized the data up to 6 months prior to participation in B7841003 for de novo participants and up to 6 months prior to participation in B7841002 for roll over participants.
Population: This efficacy analysis was conducted in the Per Protocol Analysis Set (PPAS) that included all participants who received at least 1 dose of investigational product and did not have any major protocol deviations.
Measure: Mean (Standard Deviation); unit: Bleeding episodes/participant/year
Arm/Group | Cohort 1: 300mg - 300mg Non-Inhibitor | Cohort 2: 300mg Loading + 150mg - 300mg Loading + 150mg Non-Inhibitor | Cohort 3: 450mg - 300mg Loading + 150mg Non-Inhibitor | Cohort 4: 300mg - 300mg Inhibitor | Cohort 5: De Novo 300mg Loading + 150mg Inhibitors
Number analyzed (Participants) | 5 | 4 | 4 | 5 | 2
Bleeding episodes/participant/year
  Pre-Treatment | 22.000 (7.8740) | 14.000 (1.6330) | 22.000 (13.5647) | 18.400 (1.6733) | 15.000 (4.2426)
  On-Study | 2.971 (2.7895) | 3.586 (7.1726) | 1.916 (1.4492) | 0.000 (0.0000) | 2.488 (3.5187)

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 393
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Arm/Group | Cohort 1: 300mg - 300mg Non-Inhibitor | Cohort 2: 300mg Loading + 150mg - 300mg Loading + 150mg Non-Inhibitor | Cohort 3: 450mg - 300mg Loading + 150mg Non-Inhibitor | Cohort 4: 300mg - 300mg Inhibitor | Cohort 5: De Novo 300mg Loading + 150mg Inhibitors
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4 | 0/4 | 0/5 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/4 | 0/4 | 0/5 | 0/2
Other Adverse Events (participants affected / at risk) | 5/5 | 2/4 | 4/4 | 2/5 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: 300mg - 300mg Non-Inhibitor (N=5) | Cohort 2: 300mg Loading + 150mg - 300mg Loading + 150mg Non-Inhibitor (N=4) | Cohort 3: 450mg - 300mg Loading + 150mg Non-Inhibitor (N=4) | Cohort 4: 300mg - 300mg Inhibitor (N=5) | Cohort 5: De Novo 300mg Loading + 150mg Inhibitors (N=2)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: 300mg - 300mg Non-Inhibitor (N=5) | Cohort 2: 300mg Loading + 150mg - 300mg Loading + 150mg Non-Inhibitor (N=4) | Cohort 3: 450mg - 300mg Loading + 150mg Non-Inhibitor (N=4) | Cohort 4: 300mg - 300mg Inhibitor (N=5) | Cohort 5: De Novo 300mg Loading + 150mg Inhibitors (N=2)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint warmth (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-11-08): https://cdn.clinicaltrials.gov/large-docs/21/NCT03363321/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-08): https://cdn.clinicaltrials.gov/large-docs/21/NCT03363321/SAP_001.pdf